CLINICAL TRIAL: NCT07075913
Title: Analgesic Efficacy of Adding Dexmedetomidine to Erector Spinae Plane Block Versus Subcostal Transverse Abdominis Plane Block in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Lamees Elsayed Ali Soliman Shaloof, Resident of Anesthesia, Surgical Intensive Care and Pain Therapy, Faculty of Medicine, Kafr-Elsheikh University, Kafr-Elsheikh, Egypt., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-624
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Analgesic Efficacy; Dexmedetomidine; Erector Spinae Plane Block; Subcostal Transverse Abdominis Plane Block; Laparoscopic Cholecystectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Patients received an ultrasound-guided subcostal transverse abdominis plane block with injection of 10 ml bupivacaine 0.25 %, 5ml lignocaine 2 % plus 0.5 μg/kg dexmedetomidine in a 20 ml volume.
  Interventions: Other: Subcostal transverse abdominis plane block
- Group II (Experimental): Patients will receive an ultrasound-guided erector spinae plane block (ESPB) with injection of 10 ml bupivacaine 0.25%, 5 ml lignocaine 2 % plus 0.5 μg/kg dexmedetomidine in a 20 ml volume.
  Interventions: Other: Erector spinae plane block

INTERVENTIONS:
Other: Subcostal transverse abdominis plane block — Patients received an ultrasound-guided subcostal transverse abdominis plane block with injection of 10 ml bupivacaine 0.25 %, 5ml lignocaine 2 % plus 0.5 μg/kg dexmedetomidine in a 20 ml volume.
  Arms: Group I
Other: Erector spinae plane block — Patients will receive an ultrasound-guided erector spinae plane block (ESPB) with injection of 10 ml bupivacaine 0.25%, 5 ml lignocaine 2 % plus 0.5 μg/kg dexmedetomidine in a 20 ml volume.
  Arms: Group II

SUMMARY:
Our scientific work aimed to evaluate the analgesic efficacy of dexmedetomidine as an adjuvant to erector spinae plane block versus subcostal transverse abdominis plane block in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) is the most commonly performed surgical procedure for the management of cholelithiasis. Acute pain after LC consists of somatic, parietal, and referred pain caused by trocar insertion, gall bladder resection, carbon dioxide insufflation, and other factors.

The subcostal transverse abdominis plane (SCTAP) block is the deposition of local anesthetic in the transverse abdominis plane inferior and parallel to the costal margin.

Ultrasound-guided erector spinae plane block (ESPB) is a popular, interfascial regional technique initially described for managing thoracic neuropathic pain.

Dexmedetomidine is an alpha-2 adrenergic receptor agonist that has been the focus of interest due to its sedative, analgesic, perioperative sympatholytic, and cardiovascular-stabilizing effects, resulting in reduced anesthetic requirements.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 60 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I and II.
* Patients were planned to undergo laparoscopic cholecystectomy.

Exclusion Criteria:

* Patient's refusal to participate in the study.
* ASA III, IV.
* History of clinically significant cardiac, hepatic, renal, respiratory or neurological disease.
* Coagulopathy and bleeding disorders.
* Known allergy to any drug included in the study.
* Systemic or local infection at the puncture site.
* Body mass index (BMI) >35 (kg/m2).
* Failed technique.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Total dose of morphine consumption | 24 hours postoperatively
  If the Visual analogue scale (VAS) is ≥ 3, IV morphine was given as a bolus of 2 mg (body weight < or = 60 kg) or 3 mg (body weight > 60 kg) with 5 minutes' lockout interval.

SECONDARY OUTCOMES:
Heart rate | 24 hours postoperatively
  Heart rate was recorded at baseline, after injection then every 30 minutes till the end of surgery and after surgery at 0, 2, 4, 6, 8, 12, 16 and 24 h.
Mean arterial pressure | 24 hours postoperatively
  Mean arterial pressure was recorded at baseline, after injection then every 30 minutes till the end of surgery and after surgery at 0, 2, 4, 6, 8, 12, 16 and 24 h.
Intraoperative opioid consumption | Intraoperatively
  Intraoperative opioid consumption was recorded.
Time to first rescue analgesia | 24 hours postoperatively
  Time to first rescue analgesia was recorded from the end of surgery till first dose of morphine administrated.
Degree of pain | 24 hours postoperatively
  Visual analogue scale (VAS) was assessed after surgery at 0, 2, 4, 6, 8, 12, 16, 18, and 24 h [where (0 = no pain and 10 = severe pain)].
Incidence of complications | 24 hours postoperatively
  Incidence of complications such as pneumothorax, local anesthetic systemic toxicity (LAST), bradycardia, hypotension, nausea, vomiting, and failed block were recorded.
Patient satisfaction | 24 hours postoperatively
  Degree of patient satisfaction will be assessed on a 3-point scale; (1= Unsatisfied, 2= neither satisfied nor unsatisfied, 3= satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.